CLINICAL TRIAL: NCT04171076
Title: Transcutaneous Spinal Cord Stimulation for Freezing of Gait in Parkinson Disease
Brief Title: Transcutaneous Spinal Cord Stimulation for Parkinson Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Rubens Gisbert Cury, Principal investigator, University of Sao Paulo General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USaoPauloGH 1
Record Dates: First submitted 2019-11-10; First posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Parkinson Disease; Gait, Rigid
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Intervention: non-invasive spinal cord stimulation
  Interventions: Procedure: Transcutaneous spinal cord stimulation

INTERVENTIONS:
Procedure: Transcutaneous spinal cord stimulation — Theta burst stimulation at thoracic level (T5) over 2 minutes

SUMMARY:
Spinal cord stimulation has been used to treat gait problems in Parkinson's disease, with positive results along some studies. The use of non-invasive stimulation can be an alternative to stimulate the spinal corn.

DETAILED DESCRIPTION:
Spinal cord stimulation has been used to treat gait problems in Parkinson's disease, with positive results along some studies. The use of non-invasive stimulation can be an alternative to stimulate the spinal corn. In this pilot trial, the investigators recruit participants with Parkinson' disease and freezing of gait. The aim of the study is to explore the safety along the non-invasive magnetic thoracic spinal cord stimulation as well the effect on gait problems, especially freezing of gait, prospectively, in an open-label fashion.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of advanced idiopathic Parkinson's disease
* significant freezing of gait despite optimized treatment with medications and rehabilitation program

Exclusion Criteria:

* psychiatric symptoms
* dementia
* cardiac pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — aged 18 years or higher
Enrollment: 5 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2019-11-15 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Freezing of gait score | One week
  The primary outcome is the freezing of gait score. 12-item scale, each item scores 3 points at maximum; the score ranges from 0-36; higher scores mean higher severity

SECONDARY OUTCOMES:
Gait speed | baseline, 1 week, 4 week
  Gait speed measured through the time to up and go - It uses the time that a person takes to rise from a chair, walk ten meters, turn around, walk back to the chair, and sit down.
Freezing of gait questionnaire | baseline, 1 week, 4 week
  The freezing of gait questionnaire assess the freezing of gait severity in 9-item scale ( ranging from 0-28 points); higher score mean higher severity
Safety of the intervention - urinary incontinence | 1 week, 4 week
  Incidence of Patients self report problems: urinary incontinence. The urinary incontinence will be measure through the Revised Urinary Incontinence Scale, ranging from 0 to 16. Higher scores mean higher the urinary symptoms.
Safety of the intervention - lower limb strength. | 1 week, 4 week
  Incidence of Patients self report problems: worsening in gait due to weakness. The lower limb strength will be measure through the neurologic exam. The force degree ranges from 0 - none, to 5 - normal strength.

CONTACTS AND LOCATIONS:
Locations (1):
- University of São Paulo, São Paulo, São Paulo, Brazil